CLINICAL TRIAL: NCT02181348
Title: Role of Vitamin E in Enhancing Erythropoiesis and the Molecular Mechanism of the Action of Vitamin E on Erythropoietin-secreting Cells
Brief Title: Effect of Vitamin E Supplementation on Hemoglobin Levels in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Tanveer Jilani, Senior Instructor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJilani
Record Dates: First submitted 2014-07-02; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Anemia
Keywords: Vitamin E, Hemoglobin, mild anemia
MeSH Terms: conditions — Anemia | interventions — Vitamin E; Tocopherols; Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Vitamin E supplementation) (Active Comparator): Vitamin E 400 mg once daily for 3 months
  Interventions: Drug: Vitamin E
- placebo (edible oil) (Placebo Comparator)
  Interventions: Drug: placebo (edible oil)

INTERVENTIONS:
Drug: Vitamin E — dl-alpha tocopheryl acetate 400 mg once daily for 3 months
  Other Names: Evion
  Arms: Intervention (Vitamin E supplementation)
Drug: placebo (edible oil)
  Arms: placebo (edible oil)

SUMMARY:
Anemia is one of the major health problems of the developing countries of the world [1]. According to the WHO reference criteria, an adult is labeled as anemic, if the blood hemoglobin concentration falls below 13.0 g/dL in men or less than 12.0 g/dL in the non-pregnant women [2]. Hemoglobin concentrations below the lower limit of normal are a common laboratory finding in apparently healthy people in general population all over the world [3-5]. Many of these mildly anemic individuals are not investigated sufficiently to establish the probable cause of their anemia and thus may end up with morbidity and health problems, especially the young women in developing countries [4].

Only few studies on the use of vitamin E in the correction of anemia have been published and hardly any on correction of mild anemia in healthy adults. The objective of this intervention study was to investigate the association of vitamin E supplementation with post-supplemental blood hemoglobin levels in mildly anemic healthy Pakistani adults.

DETAILED DESCRIPTION:
Anemia is one of the major health problems of the developing countries of the world [1]. According to the WHO reference criteria, an adult is labeled as anemic, if the blood hemoglobin concentration falls below 13.0 g/dL in men or less than 12.0 g/dL in the non-pregnant women [2]. Hemoglobin concentrations below the lower limit of normal are a common laboratory finding in apparently healthy people in general population all over the world [3-5]. Many of these mildly anemic individuals are not investigated sufficiently to establish the probable cause of their anemia and thus may end up with morbidity and health problems, especially the young women in developing countries [4].

A few human studies during the past few years have suggested the possible use of antioxidant vitamins in the correction of anemia [6]. Vitamin E is an essentially required lipophilic vitamin with a variety of antioxidant and non-antioxidant functions. It has been shown that treatment with vitamin E resulted in increased number of colony forming units of erythroid precursors in experimental animals and protected their bone marrow against drug- induced toxicity [7]. In some of the clinical trials in patients with hematological disorders, vitamin E supplementation showed decrease in red blood cell deformability and enhanced blood hemoglobin levels [8,9]. Although clinical benefits of vitamin E on increasing hemoglobin levels in some disease states have been published, yet its effect on a presumably healthy adult population with no abnormality other than mild anemia has hardly been reported.

Hypothesis:

Vitamin E supplementation for three months to mildly anemic healthy adults (with no past history of any iron supplements) would result into improved post-supplemental levels of blood hemoglobin compared to their basal levels.

Objective of the present study: To investigate the association of vitamin E supplementation in mildly anemic healthy adults with the post-supplemental blood hemoglobin levels in a general population of Karachi, Pakistan.

Study Participants

In this placebo-controlled and single blinded study, 357 healthy volunteer subjects, 235 males and 122 non-pregnant females of age 18-45 years were recruited and enrolled through general practitioners' (GP) clinics from various localities of Karachi and from the personnel of the Aga Khan University, Karachi. The recruitment was started in 2008 and completed in 2011. The clinical examination of study subjects was carried out by a general physician. The participants were nonsmokers; had no history of gastrointestinal disorders or chronic disease or iron deficiency during the last 6 months; had not taken vitamin E supplements or received blood transfusion during the past 6 months, and were not dehydrated. They were screened for the presence of mild anemia (10.0-13.9 g/dL, in males and 8.4-11.2 g/dL, in non-pregnant females using the criteria followed by the Aga Khan University Hospital (AKUH), Karachi.

After screening, 124 subjects (80 males and 44 females) who were found to be mildly anemic and fulfilling the criteria were included in the intervention trial. Eighty two subjects were randomly placed in Intervention group and 42 in the Control group.

Supplementation

Intervention group: Each subject was provided with 400 mg oral capsule of vitamin E (Evion, containing dl-alpha tocopheryl acetate) and was asked to take one capsule daily continuously for three months.

Control group: Each subject was provided with placebo (edible oil) capsules to be taken once daily for three consecutive months. The placebo capsules were identical to vitamin E capsules in size, shape, color, appearance and taste. The compliance of the participants was monitored by counting the number of capsules consumed after every 4 weeks.

Blood Sampling and Measurement of Biomarkers

Ten mL of fasting blood was collected before the start of supplementation from each participant and another sample (10 mL) was obtained after 3 months of supplementation. Each blood sample was divided into two equal parts; one part of blood was transferred to a tube containing anticoagulant , while the other part was transferred to a plain tube for obtaining serum. Blood samples were analyzed for blood hemoglobin levels in an automated hematology analyzer. Serum/plasma samples were kept frozen at -70 degree Centigrade for analysis of other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* mildly anemic (on the basis of screening) volunteer males and non-pregnant and non-lactating females, giving written informed consent.
* normolipidemic, normotensive
* no history of: i. diabetes, hyperlipidemia, obesity, asthma, cancer, respiratory, cardiovascular, nervous, gastrointestinal, hepatic, urogenital, musculoskeletal, endocrine, psychiatric, sexually-transmitted disease, during the last 5 years.

ii. severe acute or chronic blood loss during last 6 months. iii. bleeding or clotting abnormality during last 1 year. iv. regular cigarette smoking, tobacco chewing v. consumption of vitamin E, vitamin B12, folate, iron or antioxidant during the last 6 months prior to enrollment.

Exclusion Criteria:

* pregnant and lactating females.
* cigarette smoking, tobacco chewing, alcohol consumers
* blood transfusions during the last 1 year
* history of diabetes mellitus, hypertension, dyslipidemia , obesity asthma, cancer, respiratory, renal, nervous, gastrointestinal, hepatic, urogenital, musculoskeletal, endocrine, psychiatric, cardiovascular disorder/disease during the last five years.
* severe acute blood loss during last 6 months.
* bleeding or clotting abnormalities during the last 1 year.
* consumed vitamin E, B12, folate, iron or antioxidants supplements during the last 6 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 357 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin levels | Change in hemoglobin levels in mildly anemic adults at baseline and after 3 months of intervention (vitamin E or placebo) in all the participants in intervention arm and placebo arm (end-line).
  Hemoglobin levels in blood were determined in mildly anemic adults before intervention (baseline) and after 3 months of supplementation with vitamin E 400 mg per day (end-line).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tanveer Jilani, MBBS, M.Phil, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] 1. Milman N (2011) Ann Hematol 90:369-377. 2. WHO (2011) Vitamins and Mineral Nutrition Information System. Geneva, World Health Organization, (WHO/NMH/NHD/MNM/11.1). 2,2014) 3. Bulliyy G, Mallick G, Sethy GS, Kar SK (2007) Int J Adolesc Med Health 19(4): 395-406. 4. Kusumi E, Shoji M, Endou S, Kishi Y, Shibata T, et al. (2006) Int J Hematol 84(3): 217-219. 5. Ziauddin Hyder S, Persson LK, Chowdhury A, Ekstrom EC (2001) Public Health Nutr 4(1): 79-83. 6. Ahmed J, Zaman MM, Ali K (2003) Mymensingh Med J 12(2): 120-123. 7. Gogu SR, Lertora JJ, George WJ, Hyslop NE, Agrawal KC (1991) Exp Hematol 19: 649-652. 8. Jaja SI, Aigbe PE, Gbenebitse S, Temiye EO (2005) Niger Postgrad Med J 12: 110-114. 9. Sultana N, Begum N, Begum S, Ferdousi S, Ali T (2009) Pak J Physiol 5(1):25-28.
- [Derived] Jilani T, Azam I, Moiz B, Mehboobali N, Perwaiz Iqbal M. Positive Association of Vitamin E Supplementation with Hemoglobin Levels in Mildly Anemic Healthy Pakistani Adults. Int J Vitam Nutr Res. 2015;85(1-2):39-49. doi: 10.1024/0300-9831/a000222. PMID 26780276